CLINICAL TRIAL: NCT03079050
Title: An Open-Label Trial of Dexlansoprazole 60mg for the Relief of Heartburn During the Fasting Month of Ramadan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM.AS1.48
Record Dates: First submitted 2017-02-27; First posted 2017-03-14 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-02

CONDITIONS: GERD; Proton Pump Inhibitor
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Dexlansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 1 (Experimental): 34 patients will be assigned to take Dexlansoprazole 60mg over the 2nd, 3rd, and 4th weeks of the month of Ramadan.
  Interventions: Drug: Dexlansoprazole 60 MG

INTERVENTIONS:
Drug: Dexlansoprazole 60 MG — This drug will be given to 34 random patients during the 2nd, 3rd, and 4th weeks of the month of Ramadan to assess its ability to relieve GERD symptoms
  Other Names: Dexilant 60 MG

SUMMARY:
Dexlansoprazole modified release (MR), the R-enantiomer of Lansoprazole, is an FDA approved drug (2009) for the management of erosive esophagitis and nonerosive reflux disease 1. Dexlansoprazole has a unique dual delayed-release delivery system designed to address unmet needs that may accompany traditional proton pump inhibitors, with two separate pH-depended release phases, the first in the proximal duodenum and the second in the more distal small intestine. This dual release system extends the plasma concentration and pharmacodynamics effects beyond those of single-release PPIs, allowing for dosing at any time of the day without regard to meals 1. A study conducted by Fass et al. has shown that the use of dexlansoprazole MR 30 mg in patients with symptomatic GERD is significantly more effective than placebo in improving nocturnal heartburn, reducing GERD-related sleep disturbances, and consequently improving work productivity, sleep quality and quality of life 2.

Because of its pharmacokinetic properties, Dexlansoprazole modified release (MR) may prove beneficial in optimizing the management of GERD and the associated burdens that often surface after the heavy evening and Suhur meals, such as increased nocturnal symptoms and poor sleep quality.

DETAILED DESCRIPTION:
To investigate the efficacy and quality of life improvement of Dexlansoprazole 60mg taken once daily at Iftar time in patients with known symptomatic heartburn exacerbated in Ramadan and who are not on daily treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18-75 years old
* Fasting in Ramadan
* No daily PPI use
* Individuals willing to sign consent form
* Patients owning a smartphone and able to use a smartphone application

Exclusion Criteria:

* Known erosive GERD on PPI
* Pregnant females
* Prior gastric surgery
* Long standing diabetes mellitus (≥10 years of disease)
* Frequent NSAID use (>3x/week)
* Morbid obesity (BMI>35)
* History of recent (<6 months) upper GI bleeding
* Patients who do not own a smartphone or who cannot use a smartphone application
* Known allergy to PPIs
* Known history of poor compliance or adherence and active psychological problems which might impact adherence

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Heartburn Relief | 1 month
  The mean number of days during Ramadan with complete relief of heartburn symptoms, including nocturnal symptoms.

SECONDARY OUTCOMES:
Days with partial relief of heartburn symptoms | 1 month
  Days with partial relief of heartburn symptoms
Days with relief of nocturnal heartburn symptoms | 1 month
  Days with relief of nocturnal heartburn symptoms
Improvement in sleep qualit | 1 month
  The number of nocturnal sleeping hours will be assessed daily
Side effects/tolerability of Dexlansoprazole 30mg vs. Dexlansoprazole 60mg | 1 month
  "Side effects and tolerability" Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut - Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Behm BW, Peura DA. Dexlansoprazole MR for the management of gastroesophageal reflux disease. Expert Rev Gastroenterol Hepatol. 2011 Aug;5(4):439-45. doi: 10.1586/egh.11.37. PMID 21780890
- [Background] Fass R, Johnson DA, Orr WC, Han C, Mody R, Stern KN, Pilmer BL, Perez MC. The effect of dexlansoprazole MR on nocturnal heartburn and GERD-related sleep disturbances in patients with symptomatic GERD. Am J Gastroenterol. 2011 Mar;106(3):421-31. doi: 10.1038/ajg.2010.458. Epub 2011 Jan 11. PMID 21224838
- [Background] Fass R, Inadomi J, Han C, Mody R, O'Neil J, Perez MC. Maintenance of heartburn relief after step-down from twice-daily proton pump inhibitor to once-daily dexlansoprazole modified release. Clin Gastroenterol Hepatol. 2012 Mar;10(3):247-53. doi: 10.1016/j.cgh.2011.11.021. Epub 2011 Dec 7. PMID 22155561
- [Background] Solem C, Mody R, Stephens J, Macahilig C, Gao X. Mealtime-related dosing directions for proton-pump inhibitors in gastroesophageal reflux disease: physician knowledge, patient adherence. J Am Pharm Assoc (2003). 2014 Mar-Apr;54(2):144-53. doi: 10.1331/JAPhA.2014.13117. PMID 24632930
- [Background] Kahrilas PJ, Shaheen NJ, Vaezi MF, Hiltz SW, Black E, Modlin IM, Johnson SP, Allen J, Brill JV; American Gastroenterological Association. American Gastroenterological Association Medical Position Statement on the management of gastroesophageal reflux disease. Gastroenterology. 2008 Oct;135(4):1383-1391, 1391.e1-5. doi: 10.1053/j.gastro.2008.08.045. No abstract available. PMID 18789939
- [Background] Abbas Z. Gastrointestinal health in Ramadan with special reference to diabetes. J Pak Med Assoc. 2015 May;65(5 Suppl 1):S68-71. PMID 26013794
- [Derived] Rimmani HH, Rustom LBO, Rahal MA, Shayto RH, Chaar H, Sharara AI. Dexlansoprazole is Effective in Relieving Heartburn during the Fasting Month of Ramadan. Dig Dis. 2019;37(3):188-193. doi: 10.1159/000496091. Epub 2019 Jan 9. PMID 30625462